CLINICAL TRIAL: NCT06367114
Title: Phase Ⅱ Clinical Trial of ssCART-19 Cell Injection in the Treatment of CD19 Positive Relapsed or Refractory Acute Lymphoblastic Leukemia (Including Central Nervous System Infiltration)
Brief Title: Clinical Trial of ssCART-19 Cell Injection in the Treatment of Relapsed or Refractory Acute Lymphoblastic Leukemia (Including Central Nervous System Infiltration)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Unicar-Therapy Bio-medicine Technology Co.,Ltd (Industry)
Collaborators: The First Affiliated Hospital of Soochow University (Other); Peking University People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ssCART-19-II-1
Record Dates: First submitted 2024-04-03; First posted 2024-04-16 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Relapsed or Refractory Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Recurrence; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ssCART-19 Cells (Experimental): Route of administration: Intravenous injection.
  Lymphodepletion conditioning:
  Lymphodepletion will be conducted several days prior to ssCART-19 cells infusion.
  A combination of fludarabine and cyclophosphamide will be used for lymphodepletion.
  Interventions: Biological: ssCART-19; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: ssCART-19 — Split-Dose of ssCART-19 cells will be infused, and classic "3+3" dose escalation will be applied.
Drug: Fludarabine — Fludarabine is used for lymphodepletion.
Drug: Cyclophosphamide — Cyclophosphamide is used for lymphodepletion.

SUMMARY:
This study is a Phase II, single-arm, open-label, non-randomized, dose-escalation clinical trial to evaluate the efficacy and safety of ssCART-19 Cell Injection in the treatment of patients with CD19 positive Relapsed or Refractory acute lymphoblastic leukemia, including central nervous system infiltration.

DETAILED DESCRIPTION:
This study is a Phase II, single-arm, open-label, non-randomized, dose-escalation clinical trial to evaluate the efficacy and safety of ssCART-19 Cell Injection in the treatment of patients with CD19 positive Relapsed or Refractory acute lymphoblastic leukemia, including central nervous system infiltration. The study consists of screening period (8 weeks), treatment period (4 weeks), and follow-up period. All subjects who have received ssCART-19 infusion will be followed for safety and efficacy up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent is signed by the subject.
2. Age 18 to 65.
3. Relapsed or refractory acute lymphoblastic leukemia (ALL), According to the Chinese Guidelines for the Diagnosis and Treatment of Acute Lymphoblastic Leukemia in Adults (2021) those who need to fulfill one of the following conditions: (1)refractory leukemia: failure to reach CR/CRi after standard induction therapy (generally referred to as the 4-week regimen or Hyper-CVAD regimen). (2) Recurrence of leukemia: patients who have already reached CR have primitive cells in their peripheral blood or bone marrow (proportion>5%). (3)Patients with Ph+ ALL are eligible if they do not reach CR after at least two lines of TKI therapy or relapse after CR (except those who are intolerant to TKI therapy, have contraindications to TKI therapy or have T315i mutations). (4)Relapse after autologous or allogeneic hematopoietic stem cell transplantation(HSCT).
4. Bone marrow with ≥ 5% lymphoblasts by morphologic assessment at screening (morphological examination)
5. CD19 tumor expression demonstrated in bone marrow by flow cytometry
6. Eastern cooperative oncology group (ECOG) performance status of 0 to 1.
7. Adequate organ function at screening defined as: a.Left ventricular ejection fraction ≥ 50% by echocardiogram. b.Creatinine ≤1.5× upper limit of normal (ULN), or creatinine clearance ≥ 60 mL/min (Cockcroft and Gault). c.ALT and AST≤3×ULN, total bilirubin ≤2×ULN. d.dyspnea (CTCAE v5.0) ≤ grade 1 (shortness of breath during moderate activity) and blood oxygen saturation > 91% without oxygen inhalation as determined by investigators.
8. Vascular conditions for apheresis.
9. Females of childbearing potential who have a negative pregnancy test by blood human chorionic gonadotropin (HCG) (immunofluorescence) during the screening period and who agree to use effective contraception for at least 1 year after the infusion; male subjects whose partner is a female of childbearing potential must agree to use an effective barrier method of contraception for at least 1 year after the infusion and to refrain from sperm donation
10. The estimated survival time is more than 3 months

Exclusion Criteria:

1. Isolated extra-medullary disease relapse (except central nervous system infiltration).
2. Presence of other tumors that have not been eradicated within 5 years prior to screening that the investigator assesses may have a potential impact on the tumor.
3. Has past or at screening CNS diseases other than this disease, such as epilepsy, cerebrovascular ischemia/hemorrhage, dementia, cerebellar diseases or any CNS-related autoimmune diseases.
4. Has had treatment with any prior anti-CD19 therapy, except for leukemia cells with a positive proportion of CD19 ≥80%.
5. Therapeutic systemic doses of hormone were stopped < 72 hours prior to apheresis. However, the following physiological replacement doses of hormone are allowed: < 10 mg/day prednisone or equivalent amounts of other steroid hormones.
6. Received donor lymphocyte infusion (DLI) within 6 weeks prior to ssCART-19 infusion
7. Radiotherapy before ssCART-19 infusion:Non-CNS site of radiation completed < 2 weeks prior to ssCART-19 Infusion; CNS directed radiation completed < 8 weeks prior to ssCART-19 infusion.
8. Has had treatment with any anti-T cell antibody therapy within 4 weeks prior to monocyte collection.
9. Patients complying with any of hepatitis B surface antigen (HBsAg) and/or hepatitis B e antigen (HBeAg) positive, hepatitis B e antibody (HBe-Ab) and/or hepatitis B core antibody (HBc-Ab) positive and HBV-DNA copies being more than the lower limit of detection, hepatitis C antibody (HCV-Ab) positive, and HCV-DNA copies being more than the lower limit of detection, anti-treponemia pallidum antibody (TP-Ab) positive, human immunodeficiency virus (HIV) antibody positive, EBV-DNA, and CMV-DNA copies being more than the lower limit of detection.
10. Patients with active infections or uncontrolled infections that required systemic treatment in screening (except for mild genitourinary infections and upper respiratory infections).
11. Prior to signing the informed consent, have had cardiac angioplasty or stent placement within 12 months, or have had III-IV congestive heart failure (NYHA), or have had myocardial infarction, unstable angina, or other heart disease determined by the investigator to be ineligible for enrollment within 6 months, or QTc interval ≥480ms (QTc interval calculated by Fridericia formula) during screening, Hypertension that has not been controlled after standard treatment (systolic ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg) or pulmonary hypertension.
12. Patients have systemic diseases as judged by investigators to be unstable: including, but not limited to, severe liver, kidney, or metabolic diseases requiring medical treatment.
13. Patients with active or uncontrolled autoimmune disease, primary or secondary immunodeficiency.
14. Has had severe immediate hypersensitivity reaction to any drug to be used in this study.
15. Has had treat with live vaccine within 6 weeks prior to screening.
16. Pregnant or lactating women.
17. A history of autoimmune diseases (e. g., Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus) requiring systemic immunosuppressive/systemic disease modifying medications within the past 2 years
18. Patients with a history of allogeneic hematopoietic stem cell transplantation within 12 weeks prior to apheresis, acute graft-versus-host disease (GVHD) or moderate to severe chronic GVHD within 4 weeks prior to screening; Patients who received systemic drug therapy for GVHD within 4 weeks prior to infusion.
19. Participating in any other study and have received any other investigational drug within 4 weeks prior to screening.
20. Patients with other conditions making the patients unsuitable for this study as judged by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Determine the efficacy of ssCART-19 cells in patients with CD19-positive relapsed or refractory acute B lymphoblastic leukemia (r/r B-ALL). | At 3 months after infusion
  Overall Remission Rate (ORR), which includes Complete Remission (CR) and complete remission with partial hematologic recovery (CRh) and Complete Remission with Incomplete Blood Count Recovery (CRi) as determined by Independent Review Committee (IRC).

SECONDARY OUTCOMES:
Observe the anti-tumor response of ssCART-19 cells to refractory or relapsed acute lymphoblastic leukemia. | 3 months
  Overall remission rate (ORR) with negative micro residual disease (MRD) within 3 months after ssCART-19 infusion.
Best overall response (BOR)assessment during the 3 months after ssCART-19 infusion. | 3 months
  The proportion of patients who have achieved the best effect (CR or CRi) after the experimental treatment.
Duration of response (DOR) | 24 months
  DOR means the duration from reaching the response CR or CRi to the first defined relapse, or death due to any cause, whichever comes first.
Recurrence free survival (RFS) | 24 months
  RFS means the duration from reaching the response CR or CRi to the first defined relapse, or death due to any cause, whichever comes first.
Event Free Survival (EFS) | 24 months
  EFS means duration from the ssCART-19 Cell Injection infusion to death for any reason after remission, relapse, treatment failure, no response, or termination (because of death, adverse event, lack of efficacy, progression, new anti-tumor treatments.
Overall survival (OS) | 24 months
  OS is defined as the time from the ssCART-19 Cell Injection infusion to the date of death due to any cause.
Incidence of adverse events following ssCART-19 infusion | 24 months
  Therapy-related adverse events were recorded and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0) Dose-limiting toxicity after ssCART-19 infusion.
Pharmacodynamic of ssCART-19 cells | 28 days
  Peak value of eripheral blood (Cmax)
Pharmacodynamic of ssCART-19 cells | 28 days
  Area under the eripheral blood concentration versus time curve (AUC)
Pharmacodynamic of ssCART-19 cells | 28 days
  Time of peak value

OTHER OUTCOMES:
Anti-drug antibody | 24 months
  Detect titer of anti-drug antibody (ADA)

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Shanghai Unicar-Therapy Bio-medicine Technology Co., Ltd., Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Soochow University, Suzhou